CLINICAL TRIAL: NCT00738088
Title: The Use of Glycaemic Response to Sulphonylureas as a Tool to Investigate Type 2 Diabetes Pathophysiology
Brief Title: Variation in Sulphonylurea Response in Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Following Regulator inspection in 2009, study terminated as inadequate approvals were in place
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Ewan Pearson, Professor of Diabetic Medicine, NHS Tayside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007DM02; EudraCT 2007-000594-29
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Sulphonylurea; Pharmacogenetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Withdrawal of sulphonylurea for 6 weeks, then re-introduction for 6 weeks, assessed by fasting glucose and HbA1c
  Interventions: Drug: gliclazide

INTERVENTIONS:
Drug: gliclazide — Gliclazide 80mg bd for 6 weeks
  Other Names: Diamicron

SUMMARY:
The study hypothesis is that people who respond well to sulphonylureas have a different underlying cause for their diabetes than people who respond poorly to this medication. We are using two approaches to study this. In one approach we look at people who have previously responded well or poorly, confirm this by rechallenging them with a sulphonylurea drug, and then looking at how well they produce insulin in response to glucose and an intravenous sulphonylurea called tolbutamide. The second approach identifies people with a certain genetic predisposition to diabetes (due to changes in the TCF7L2 gene) and then looks at how well they respond to sulphonylurea medication.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age >35 and < 70
* Age of diabetes diagnosis >35 and <70
* White European
* Pre-SU HbA1c <=10%
* HbA1c (on treatment) <= 9%
* No myocardial infarction or Acute coronary syndrome in previous year
* No stroke or transient ischaemic attack in previous year
* No or stable (background) retinopathy (no unscheduled laser treatment in the last 6 months)
* eGFR > 60mls/min
* No Proteinuria >30mg/dl on multistix 10SG
* No active foot ulceration or infection
* Liver ALT ≤ twice the upper limit of the reference range
* Contactable by telephone

Exclusion Criteria:

* Type 1 diabetes
* HbA1c >10% prior to commencing SU
* HbA1c>9% on SU treatment
* Recent MI or Stroke within last 12 months
* Pre-proliferative or proliferative retinopathy
* eGFR<60 ml/min
* Proteinuria >30mg/dl on multistix 10SG
* Active foot ulceration or infection
* Liver ALT > twice the upper limit of the reference range
* Female planning to conceive within the study period
* Any other significant medical reason for exclusion as determined by the investigator

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2011-03-03 (Actual); Study Completion 2011-03-03 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction | 6 weeks

SECONDARY OUTCOMES:
insulin secretory response to glucose and tolbutamide | acute

CONTACTS AND LOCATIONS:
Overall Officials: Ewan R Pearson, Principal Investigator — NHS Tayside
Locations (1):
- NHS Tayside, Dundee, United Kingdom